CLINICAL TRIAL: NCT04561817
Title: An Open Label Phase II Study to Evaluate the Safety and Efficacy of Ipatasertib (GDC-0068) in Combination With Paclitaxel in Platinum-resistant Recurrent Epithelial Ovarian Cancer
Brief Title: To Evaluate the Safety and Efficacy of Ipatasertib (GDC-0068) in Combination With Paclitaxel in Platinum-resistant Recurrent Epithelial Ovarian Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Evolving data with Ipatasertib that changes the known risk / benefit background in pursuing future studies.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Amy Tiersten, Professor - Hematology Oncology, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 19-2707
Record Dates: First submitted 2020-09-08; First posted 2020-09-24 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Ovarian Neoplasms
Keywords: Platinum-resistant; Ovarian cancer; Ipatasertib; Paclitaxel; Recurrent
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — ipatasertib; Paclitaxel

STUDY DESIGN:
Intervention Model Description: For non-altered patients- An interim analysis is scheduled when the number of enrolled patients reaches 14. The research team will stop the trial for futility if 2 or less than 2 patients respond. When the total number of patients reaches the maximum sample size of 25, the research team will reject the null hypothesis and conclude that the treatment is promising if the number of responses are greater than 6; otherwise the research team will conclude that the treatment is not promising.
  For altered patients-An interim analysis is scheduled when the number of enrolled patients reaches 8. The research team will stop the entire trial of two cohorts for futility if 1 or less than 1 patients respond. When the total number of patients reaches the maximum sample size of 14, the research team will reject the null hypothesis and conclude that the treatment is promising
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PI3K/AKT mutations (altered) (Active Comparator): Participants with recurrent epithelial ovarian cancer with PI3K/AKT mutations (altered)
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel
- Without PI3K/AKT mutations (non-altered) (Active Comparator): Participants with recurrent epithelial ovarian cancer without PI3K/AKT mutations (non-altered)
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Ipatasertib — 400mg PO daily: day 1-21 of 28 day cycle
  Other Names: GDC-0068
Drug: Paclitaxel — 80 mg/m2 IV weekly: day 1, 8, 15 of 28 day cycle

SUMMARY:
This is a phase II open label, non-randomized, study to evaluate the safety and efficacy of Ipatasertib (GDC-0068) in combination with paclitaxel in platinum-resistant recurrent epithelial ovarian cancer.

DETAILED DESCRIPTION:
This is a phase II open label, non-randomized, study to evaluate the safety and efficacy of Ipatasertib (GDC-0068) in combination with paclitaxel in platinum-resistant recurrent epithelial ovarian cancer.

The primary objective of the study is to determine - the safety and objective response rate of treatment with ipatasertib (GDC-0068) in combination with paclitaxel in platinum-resistant recurrent epithelial ovarian cancer at week 12 for two cohorts of patients: with PI3K/AKT mutations (altered) and without PI3K/AKT mutations (non-altered)

About 39 patients will participate in the study and the accrual will take place over a course of 30 months Patients will be treated until disease progression and followed for 1 year thereafter.

The two drugs are ipatasertib and paclitaxel.

* Ipatasertib will be given 400mg PO daily: day 1-21 of 28 day cycle
* Paclitaxel will be given 80mg/m2 IV weekly: day 1, 8, 15 of 28 day cycle

The study hypothesis is that the combination of Ipatasertib (GDC-0068) plus paclitaxel will safely induce a tumor response and increase the objective response rate in patients with platinum-resistant recurrent epithelial ovarian cancer, with or without PI3K/AKT mutations.

This trial will enroll patients with platinum-resistant recurrent epithelial ovarian cancer. Given the relatively poor prognosis and limited treatment options for these patients, this population is considered appropriate for trials of novel therapeutic candidates. The benefit-risk ratio for ipatasertib in combination with paclitaxel is expected to be acceptable in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses

  o If a patient declines to participate in any voluntary exploratory research and/or genetic component of the study, there will be no penalty or loss of benefit to the patient and he/she will not be excluded from other aspects of the study
* Aged at least 18 years at time of signing informed consent
* A pathologic (histology or cytology) confirmed diagnosis of epithelial ovarian cancer, including fallopian or primary peritoneal cancer

  o low grade serous histology is excluded
* Radiographic evidence of recurrent epithelial ovarian cancer (ovarian, fallopian tube, or primary peritoneal cancer) that has become "platinum-resistant," defined as progression of disease within 6 months from the last dose of platinum-based chemotherapy, or platinum refractory
* Not a candidate for cytoreductive surgery
* Measurable disease (at least one lesion that can be accurately assessed repeatedly by CT or MRI) as evidenced on pre-treatment baseline CT of Chest/Abdomen/Pelvis, MRI, or PET/CT, or evaluable disease (defined as anything non-measurable- pleural effusions, lesions <1cm, etc).
* World Health Organization (WHO) performance status 0-1 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks
* Up to 3 lines of prior cytotoxic chemotherapy
* Previously received bevacizumab
* Has not received weekly paclitaxel-containing regimen, EXCEPT for in the front-line setting

  o Patients with prior paclitaxel reactions may be enrolled if they have been successfully re-treated with steroid pre-medication in the past
* Patients must use adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing (within 7 days) if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  * Post-menopausal defined as aged more than 50 years and amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 28 days after the last dose of study treatment. Women must refrain from donating eggs during this same period.

Exclusion Criteria:

* Treatment with any of the following:

  * Any investigational agents or study drugs from a previous clinical study within 28 days of the first dose of study treatment
  * Any other chemotherapy, immunotherapy or anticancer agents within 14 days of the first dose of study treatment
  * Potent inhibitors or inducers or substrates of CYP3A4 or substrates of CYP2D6 within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort)
  * Any prior exposure to Ipatasertib
* Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment
* Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study treatment
* With the exception of alopecia, any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment
* Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids for at least 2 weeks prior to start of study treatment
* Concurrent use of endocrine therapy
* As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
* Any of the following cardiac criteria:

  * Any clinically important abnormalities in rhythm, known prolonged QTc, conduction or morphology of resting ECG, complete left bundle branch block, third degree heart block
  * Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure NYHA Grade 2 or greater
  * Uncontrolled hypotension - Systolic BP <90mmHg and/or diastolic BP <50mmHg
  * Left ventricular ejection fraction (LVEF) below lower limit of normal for site
* Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

  * Absolute neutrophil count < 1.5 x 109/L
  * Platelet count < 100 x 109/L
  * Hemoglobin < 9 g/L
  * Alanine aminotransferase > 2.5 times the upper limit of normal (ULN)
  * Aspartate aminotransferase > 2.5 times ULN
  * Total bilirubin > 1.5 times ULN
  * Creatinine >1.5 times ULN concurrent with creatinine clearance < 50 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is > 1.5 times ULN
  * Proteinuria 3+ on dipstick analysis or >500mg/24 hours
  * Sodium or potassium outside normal reference range for site
* Peripheral neuropathy grade 2 or greater
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption Ipatasertib
* History of hypersensitivity to Ipatasertib, or drugs with a similar chemical structure or class to Ipatasertib
* Clinically significant abnormalities of glucose metabolism as defined by any of the following:

  * Diagnosis of type I or type II diabetes mellitus requiring insulin
  * A baseline fasting glucose value of ≥ 200 mg/dL (fasting glucose value to be obtained only if non-fasting glucose >200mg/dL)
  * Glycosylated hemoglobin (HbA1C) >7.5%
* Uncontrolled pleural effusion, pericardial effusion, or ascites
* Other malignancies within the past 3 years, with the exception of adequately resected basal or squamous carcinoma of the skin
* Clinically significant pulmonary symptoms or disease
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — A female with confirmed diagnosis of epithelial ovarian cancer, including fallopian or primary peritoneal cancer
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At the end of Cycle 1 (each cycle is 28 days)
  ORR will be measured by the percentage of patients whose cancer decreases in size on assessment. This will be measured as the sum of complete response and partial response.
Objective response rate (ORR) | At the end of Cycle 2 (each cycle is 28 days)
  ORR will be measured by the percentage of patients whose cancer decreases in size on assessment. This will be measured as the sum of complete response and partial response.
Objective response rate (ORR) | At the end of Cycle 3 (each cycle is 28 days)
  ORR will be measured by the percentage of patients whose cancer decreases in size on assessment. This will be measured as the sum of complete response and partial response.

SECONDARY OUTCOMES:
Progression free survival (PFS) | At the end of Cycle 1 (each cycle is 28 days)
  Disease status will be assessed with comprehensive radiographic studies every 3 treatment cycles (12 weeks +/- 1 week), but the development of new signs or symptoms of disease in between scheduled evaluations may prompt off-schedule radiographic or non-radiographic evaluations. Disease status will be assessed based on RECIST 1.1 criteria for measurable and non-measurable disease.
Progression free survival (PFS) | At the end of Cycle 2 (each cycle is 28 days)
  Disease status will be assessed with comprehensive radiographic studies every 3 treatment cycles (12 weeks +/- 1 week), but the development of new signs or symptoms of disease in between scheduled evaluations may prompt off-schedule radiographic or non-radiographic evaluations. Disease status will be assessed based on RECIST 1.1 criteria for measurable and non-measurable disease.
Progression free survival (PFS) | At the end of Cycle 3 (each cycle is 28 days)
  Disease status will be assessed with comprehensive radiographic studies every 3 treatment cycles (12 weeks +/- 1 week), but the development of new signs or symptoms of disease in between scheduled evaluations may prompt off-schedule radiographic or non-radiographic evaluations. Disease status will be assessed based on RECIST 1.1 criteria for measurable and non-measurable disease.
Disease control rate (DCR) | average 24 weeks
  DCR will be measured by the percentage of patients whose cancer decreases in size or remains stable over the duration of the study. This will be measured as the sum of complete response, partial response, and stable disease for greater than or equal to 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tiersten, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Dubin Breast Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee (%8Dlearned intermediary%8E) identified for this purpose.To achieve aims in the approved proposal.information on Availability of data will be provided later